CLINICAL TRIAL: NCT00208195
Title: Depakote ER Therapy for Mania Comorbid With Substance Abuse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Syed Pirzada Sattar, M.D., Creighton University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-13258
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Bipolar Disorder; Mania; Substance Abuse; Substance Dependence
Keywords: Bipolar Disorder; Mania; Substance Abuse; Substance Dependence; Comorbid
MeSH Terms: conditions — Bipolar Disorder; Mania; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Divalproex ER

SUMMARY:
The purpose of this study is to ascertain whether Depakote ER (Divalproex ER) has efficacy in the treatment of patients with bipolar disorder in the manic phase, who also have comorbid substance abuse diagnoses. It is proposed that Depakote ER will decrease scores on the Young Mania Rating Scale and the Substance Abuse Time Line Follow Back.

DETAILED DESCRIPTION:
This study will be performed in male and female subjects with a diagnosis of bipolar disorder in the manic phase of the illness who also have a comorbid diagnosis of substance abuse. This population is selected so the efficacy of Depakote ER in this population can be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 19 - 65.
2. Diagnosis of mania with comorbid substance confirmed by Structured Clinical Interview for DSM-IV.
3. Comorbid diagnoses of anxiety and/or personality disorders are permitted.
4. Ability to provide signed informed consent.
5. Stable general medical health.
6. Ability to attend outpatient research clinic.

Exclusion Criteria:

1. Dangerous to self or others.
2. Pregnancy, inability or unwillingness to use approved methods of birth control.
3. Inability or unwillingness to provide signed informed consent.
4. Diagnosis of schizophrenia, major depressive disorder.
5. Inability to attend outpatient research clinic.
6. Medical conditions, which would preclude use of Depakote.
7. Need for ongoing treatment with medication other than Depakote ER, such as antipsychotic medication.
8. Medical instability defined as likelihood of needing to change prescription medication during the course of the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-03; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures will consist of the total score on the YMRS, and the number of days abstinent from substances of abuse with the TLFB. | Patients will be evaluated on a weekly basis for the first month, then every 2 weeks for the next 2 months, then monthly for the next 3 months for a total study duration of 6 months

SECONDARY OUTCOMES:
The Addiction Severity Index (ASI), Penn Alcohol Craving Scale, and Clinical Global Impression (CGI). | Patients will be evaluated on a weekly basis for the first month, then every 2 weeks for the next 2 months, then monthly for the next 3 months, for a total study duration of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pirzada Sattar, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Psychiatry Research Center, Omaha, Nebraska, United States